CLINICAL TRIAL: NCT01599299
Title: Comparison of the Diameter, Cross-sectional Area and Position of the Left and Right Internal Jugular Vein in Adults Using Ultrasound
Brief Title: Comparison of the Right and Left Internal Jugular Vein Using Ultrasound
Status: Completed | Type: Observational
Sponsor: Catharina Ziekenhuis Eindhoven (Other)
Responsible Party: Principal Investigator, Michiel Bos, MD, Catharina Ziekenhuis Eindhoven
Other Study IDs: 1.2.2012
Record Dates: First submitted 2012-05-14; First posted 2012-05-16 (Estimated); Last update posted 2014-03-06 (Estimated); Status verified 2014-03

CONDITIONS: Comparison of the Right and Left Internal Jugular Vein Using Ultrasound
Keywords: ultrasound; left and right jugular vein; comparison

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Ultrasound, internal jugular vein: All patients who will need a central venous access (into the right jugular vein) preoperative are included.

SUMMARY:
The purpose of this study is to determine whether there is a difference between the diameter, and the cross-sectional area of the right internal in left internal jugular vein in preoperative, mechanically ventilated patients.

Secondary the relationship between the internal jugular vein to the common carotid artery will be examined.

DETAILED DESCRIPTION:
Placement of a central venous catheter (CVC) for surgery is used for hemodynamic monitoring and venous access. Most often the right internal jugular vein (RIJV) is used. The RIJV is preferred over the left-sided internal jugular vein (LIJV) because cannulation of the LIJV is more difficult and associated with a higher complication rate(1). A possible explanation for the higher complication rate can be explained by the difference in diameter between the RIJV and the LIJV. It has been demonstrated that large vessels are easier to catheterize than small ones.

Data suggest that the internal jugular veins are most often asymmetric but data are limited. Until now, there is one small prospective study in which 80 ICU patients where examined (30 patients were mechanically ventilated) which showed an asymmetry in 62,5% and a dominant RIJV in 68% and a smaller study performed by Lobato and colleagues in which 50 healthy patients were examined. They measured the cross-sectional areas of the internal jugular veins. They showed that in 80% the RIJV was greater than the LIJV. Two CT studies has been done so far. In 2009 Tartière and colleagues carried out an observational study in 190 patients. All patients were in the supine position, neutral head position an spontaneous breathing. During the CT patients were asked to hold there breath. The study showed that the diameter and cross-sectional area of the RIJV were significantly greater than those of the LIJV. A smaller retrospective CT-study (88 patients) performed by Lim et al in 2006 showed a larger RIJV in 79,5% compared to the LIJV.

Until now, there are no data known about the difference between the RIJV and LIJV in preoperative mechanical ventilated patients when ultrasound is used.

ELIGIBILITY:
Inclusion Criteria:

* all patients who will need a central venous access preoperative are included (e.g. for medication, nutrition, antibiotics)and are mechanically ventilated

Exclusion Criteria:

* < 18 years of age
* neck or head surgery in the past
* radiation therapy of the neck
* known thyroid pathology
* skeletal deformities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who will need a central venous access (into the right jugular vein) preoperative are included
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2012-03; Primary Completion 2012-06 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Comparison of the diameter, cross-sectional area and position of the left and right internal jugular vein in adults using ultrasound | Measurements are made after the patient is intubated and ventilated, prior to the surgical procedure starts.
  Comparison of the cross-sectional area and diameter of the left internal jugular vein and the right internal jugular vein

SECONDARY OUTCOMES:
Comparison of the diameter, cross-sectional area and position of the left and right internal jugular vein in adults using ultrasound | Measurements are made after the patient is intubated and ventilated, prior to the surgical procedure starts.
  The localisation of the right/left internal jugular vein in relation to the carotid artery.

CONTACTS AND LOCATIONS:
Locations (1):
- Catharina Hospital, Eindhoven, North Brabant, Netherlands